CLINICAL TRIAL: NCT03033836
Title: Pilot Study of Dolutegravir Plus Tenofovir/Lamivudine or Emtricitabine in HIV-1 Infected Transgender Women
Brief Title: Dolutegravir Plus Tenofovir/Lamivudine or Emtricitabine in HIV-1 Infected Transgender Women
Acronym: TRANSViiV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Huésped (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Principal Investigator, Omar Sued, PhD, Fundación Huésped
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FH-17
Record Dates: First submitted 2016-08-18; First posted 2017-01-27 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: HIV Infections
Keywords: transgender women
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Single Group receiving the same intervention, to evaluate retention at 48 weeks
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm (Experimental): ARV treatment based on Dolutegravir Plus Tenofovir/Lamivudine or Emtricitabine
  Interventions: Drug: ARV treatment

INTERVENTIONS:
Drug: ARV treatment — Dolutegravir 50 mg QD plus co-formulated emtricitabine 200 mg/tenofovir 300 mg QD.
  Other Names: tivicay-truvada

SUMMARY:
Prospective, open, single-arm trial of dolutegravir-tenofovir and emtricitabine or lamivudine (DTG-TDF-FTC or 3TC) in antiretroviral (ART) naïve HIV transgender women (TGW).

The primary objective of this pilot study is to determine the retention in care of TGW treated with DTG-TDF-FTC or 3TC

Secondary objectives:

* To evaluate the efficacy of the antiretroviral regimen at week 48 ;
* To describe the safety and tolerability of this regimen;
* To evaluate adherence across 48 weeks;
* To determine the patient satisfaction with this regimen;
* To identify individual, social and contextual factors associated with adherence and retention.

DETAILED DESCRIPTION:
The primary objective of this pilot study is to determine the retention in care of TGW treated with DTG-TDF-FTC.

The primary objective will be assessed by the proportion of individuals that provide information on ART use and virological outcomes at the end of the study:

* Retention under care: Proportion of enrolled and dosed individuals that provide clinical information up to 48 weeks of follow up.
* Retention on treatment: Proportion of enrolled and dosed individuals that receive study drugs up to 48 weeks of follow up.

Secondary objectives:

* To evaluate the efficacy of the antiretroviral regimen at week 48 ;
* To describe the safety and tolerability of this regimen;
* To evaluate adherence across 48 weeks;
* To determine the patient satisfaction with this regimen;
* To identify individual, social and contextual factors associated with adherence and retention.

The secondary objectives will be evaluated using the following endpoints:

1. Proportion of patients with HIV-1 RNA levels of less than 50 copies/mL at 48 weeks of treatment by the IIT-exposed snapshot FDA algorithm;
2. Frequency, type and severity of adverse events and laboratory abnormalities;
3. Pill count, analogue visual scale for adherence in each visit;
4. Changes in the scores of stigma and discrimination scales , quality of life, social support and anxiety and depression (BERGER, WBI,DUKE,CES-D,STAI) at bsl, 4,24, and 48 weeks e;.Changes in the score scales of sexual behaviors, use of drug /alcohol at bsl and at each visit .

f. Through association of baseline individual, social and contextual characteristics with percentage of adherence and retention at 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 positive serology by at least two different serological tests (rapid test, ELISA, Western Blot) or a viral load higher than 3,000 copies/mL.
2. 18 years and older.
3. Self-identified as TGW
4. ART naïve.
5. Written informed consent provided.

Exclusion Criteria:

1. Genotypic resistance to TDF and/or FTC as per IAS-USA resistance panel 2013.
2. Alcohol or drug use that might affect adherence.
3. Concomitant use of lipid-lowering drugs, interferon, interleukin-2, cytotoxic chemotherapy, dofetilide (or pilsicainide) or immunosuppressors, antacids drugs containing Ca++ and or Mg++ at study entry.
4. Opportunistic infection (CDC "C" category) or other disease and/or clinical conditions that, in the investigator's opinion, would compromise the patient's safety or outcome of the study; including malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or non-invasive cutaneous squamous cell carcinoma, or cervical intraepithelial neoplasia.
5. Treatment with any of the following agents within 28 days of screening: radiation therapy; cytotoxic chemotherapeutic agents; any immunomodulators that alter immune responses or treatment with an HIV-1 immunotherapeutic vaccine within 90 days of screening or exposure to an experimental drug or experimental vaccine within either 28 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to the first dose of the investigational product.
6. Contraindication to any of the study drugs (history of renal diseases, lab abnormalities grade 4 or any other clinical condition prior therapy that, in the opinion of the investigator, would make the subject unsuitable for the study or unable to comply with the dosing requirements).
7. Anticipated need for Hepatitis C virus (HCV) therapy during the study.
8. Creatinine clearance of <50 mL/min via Cockroft-Gault method.
9. Subjects with moderate to severe hepatic impairment (Class B or greater) as determined by Child-Pugh classification.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-12; Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Proportion of transgender women retained in care at week 48 | 48 weeks
  Proportion of enrolled and dosed individuals that complete protocol defined visits during 48 weeks of follow up.
  Retention under care: Proportion of enrolled and dosed individuals that provide clinical information up to 48 weeks of follow up.
  Retention on treatment: Proportion of enrolled and dosed individuals that receive study drugs up to 48 weeks of follow up.

SECONDARY OUTCOMES:
Proportion of individuals with HIV RNA undetectable at week 48 | 48 weeks
  Proportion of patients with HIV-1 RNA levels less than 50 copies/mL at week 48 weeks of treatment by the IIT-exposed snapshot FDA algorithm;
Percentage of Participants Experiencing Any Treatment-Emergent Laboratory Abnormality | From baseline to week 48
  Treatment-emergent laboratory abnormalities were defined as values that increase at least one toxicity grade from baseline. The most severe graded abnormality from all tests was counted for each participant.
Percentage of Participants Experiencing Treatment-Emergent Adverse Events | From baseline to week 48
  Adverse events (AEs) occurring during treatment and for 30 days following the last dose of study drug were summarized across the participant population. A participant was counted once if they had a qualifying event.
Adherence using ACTG form | From baseline to week 48
  ACTG self report adherence form will be used for baseline and follow up visits
Adherence using analogue visual scale | From week 4 to week 48
  Analogue visual scale (0-10) will be used at each follow up visit
Adherence by pill count | From week 4 to week 48
  Pill count of dispensed drugs
Quality of life by QoL Socre and Well being index | From baseline to week 48
  Changes in the scores of quality of life, will be done through Well-being Index questionnaire, this instrument will be administered to patients at baseline, week 4, 24 and week 48 .
Patient´s satisfaction with this regimen | From baseline to week 48
  Changes in the scores of social support,will be done through Duke UNC questionnaire, this instrument will be administered to patients at baseline, week 4, 24 and week 48 .

CONTACTS AND LOCATIONS:
Overall Officials: Omar Sued, MD, PhMD, Principal Investigator — Fundacion Huesped
Locations (1):
- Fundacion Huesped, Ciudad de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Yes
to publish study results